CLINICAL TRIAL: NCT03852914
Title: Prospective, Multicentre Study to Evaluate the Efficacy and Safety of Intraarticular Sodium Hyaluronate Single Injection in Patients Suffering From Osteoarthritis of the Knee
Brief Title: Efficacy and Safety of Intraarticular Sodium Hyaluronate Single Injection in Patients With Osteoarthritis of the Knee
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tedec-Meiji Farma, S.A. (Industry)
Collaborators: Alpha Bioresearch S.L. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TM-SH2%/301
Record Dates: First submitted 2019-02-22; First posted 2019-02-25 (Actual); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Sodium Hyaluronate 2% (Experimental): Each patient will receive a single injection of SH2%
  Interventions: Device: Sodium hyaluronate 2%

INTERVENTIONS:
Device: Sodium hyaluronate 2% — Each patient will receive a single injection of SH 2% and will be followed for 6 months. At 6 months follow up visit patients could be offered a second injection whenever and when they comply with the criteria established for re-treatment and will be followed for additional 6 months.

SUMMARY:
A Phase III, prospective, multicentre, non-controlled, with consecutive participant enrollment in order to evaluate the efficacy, safety and duration of the effects of the viscosupplementation with a preparation of sodium hyaluronate 2% (SH2%) from Tedec-Meiji Farma S.A. over 12 months. Adult patients diagnosed with primary osteoarthritis of the knee according to American College of Rheumatology (ACR) criteria with radiological grades II and III according to Kellgren-Lawrence scale (KL) will receive a single injection of SH2% and will be followed for 1 year with follow up visits at 6 and 12 months.

At 6 months patients could be offered a second injection whenever and when they comply with the criteria established for re-treatment and will be followed for additional 6 months

DETAILED DESCRIPTION:
Prospective, multicentre and non-controlled study. Each patient will receive a single injection of SH 2% and will be followed for 1 year with follow up visits at 6 and 12 months At 6 months follow up visit patients will be offered a second injection whenever and when they comply with the criteria established for re-treatment and will be followed for additional 6 months From the pre-inclusion V0 up to the V1 (beginning of treatment), there will be a wash-out period of 2 weeks during which only paracetamol will be allowed for osteoarthritis (OA) pain relief (maximum dose allowed:3g/day).

Paracetamol will be discontinued at least 24h before follow up visits (Treatment administration, 6 months of follow up and 12 months of follow up).

Clinical evaluation will be done every visits through VAS, WOMAC and Patient's Global Assessment/ Investigator's Global Assessment (PGA/IGA)

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 45 years of age of either sex.
* Primary knee OA of the medial or lateral femoro-tibial compartment documented according to ACR criteria with symptoms, at screening, from at least 3 months.
* KL radiological grade 2-3.
* Antero-posterior view X-Ray image of the target knee
* Pain intensity at screening in the target knee ≥40 mm and <80 mm measured by Visual Analogue Scale (VAS), and ≤ 20 mm in the contralateral knee.
* Able to understand and willing to comply with study procedures.
* Able to provide informed consent.

Exclusion Criteria:

* BMI ≥ 30 kg/m2.
* Pregnant or lactating women. Women of child-bearing age not using effective contraception.
* Severe inflammation of the target knee.
* Previous surgery in the target knee, including arthroscopy.
* Subjects with any musculoskeletal condition affecting the target knee that would impair the proper evaluation
* Patients with joint inflammatory disease, microcrystalline arthropathies and significant osteoarthritis symptoms in other joints apart from the knee, and which require pharmacological treatment.
* Underlying disease considered by the investigator that might interfere with the development and evaluation study.
* Subjects with venous or lymphatic stasis in the relevant limb.
* Previous administration of any of the following treatments: hyaluronic acid i.a. (last year); steroids i.a. or joint lavage (last 3 months), glucosamine sulfate, chondroitin sulfate or diacerein (last 3 months), NSAIDs (last 14 days), any investigational drug (last month) or its administration during this study.
* Pain in other parts of the body greater than the knee pain that could interfere with the evaluation.
* Any pathology that, under investigator judgement, interfere with the administration or assessment.
* Patients with known hypersensitivity to SH or paracetamol.
* Patients in waiting list for surgery.
* Patients awaiting disablement assessment.
* Previous participation in this protocol

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Estimated)
Dates: Start 2019-01-17 (Actual); Primary Completion 2019-10 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Change in pain intensity according to VAS (0-100mm) | 6 and 12 months after treatment
  The VAS to be used in the study consists of a horizontal line marked from 0 to 100 mm, where 0 means no pain and 100 is the greatest possible pain. Patients must draw a vertical line at the point that they believe that represents the pain intensity at that time.

SECONDARY OUTCOMES:
Change in function from baseline in the target knee | 6 and 12 months after treatment
  Physical function will be measured by using the function subscale of the Western Ontario & McMaster Universities Osteoarthritis Index (WOMAC). This index contains 24 items on different activities of daily life grouped in three subscales: pain (5 items), stiffness (2 items), and functional capacity (17 items). For each item a horizontal visual analogue scale of 0 to 100 mm with end descriptors is used, whose path goes from no pain, no stiffness, no difficulty to extreme pain, extreme stiffness, extreme difficulty.
Change in function from baseline in the target knee | 6 and 12 months after treatment
  Physical function will be measured by using the function subscale of the Western Ontario & McMaster Universities Osteoarthritis Index (WOMAC). This subscale contains 24 items on different activities of daily life grouped in three dimensions: pain, stiffness, and functional capacity. For each item a horizontal visual analogue scale of 0 to 100 mm with end descriptors is used, whose path goes from no pain, no stiffness, no difficulty to extreme pain, extreme stiffness, extreme difficulty function subscale
Percentage of patients achieving the Minimally Clinical Important Improvement (MCII) | 6 and 12 months after treatment
  The MCII is the smallest change in measurement that signifies an important improvement in a patient's symptom
Percentage of patients achieving the Patient Acceptable Symptoms State (PASS) | 6 and 12 months after treatment
  Defined as the value beyond which patients consider themselves well. According to the literature the recommended value for PASS (measured on 0-100 VAS) is < 40.
Patient and investigator global assessments | 6 and 12 months after treatment
  Both will be measured using a 5-point Likert scale. This is a five-level classification scale (0= Better, 1 = best, 2 = same, 3 = worst, 4 = much worse)

CONTACTS AND LOCATIONS:
Overall Officials: Mercedes Gimeno, PhD, Study Chair — Tedec Meiji; Carlos Gavin, PhD, Principal Investigator — Hospital Uiversitario Fundacion Alcorcón
Locations (10):
- Spain (10):
  - Hospital General de Elche, Elche, Alicánte
  - Hospital de la Marina Baixa de Villajoyosa, Villajoyosa, Alicánte
  - Hospital Universitario Fundación Alcorcón, Alcorcón, Madrid
  - Complejo Hospitalario La Coruña, A Coruña
  - Hospital Universitario Reina Sofia, Córdoba
  - Clinica Universitaria de Navarra, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid

REFERENCES:
- [Derived] Gavin C, J Blanco F, L Pablos J, Caracuel MA, Rosas J, Gomez-Barrena E, Navarro F, Coronel MP, Gimeno M. One-Year, Efficacy and Safety Open Label Study, with a Single Injection of a New Hyaluronan for Knee OA: The SOYA Trial. J Pain Res. 2021 Jul 21;14:2229-2237. doi: 10.2147/JPR.S321841. eCollection 2021. PMID 34321921